CLINICAL TRIAL: NCT05282927
Title: Implementing a Group Physical Therapy Program for Veterans With Knee Osteoarthritis: Function QUERI 2.0 (QUE 20-023)
Brief Title: Implementing Group Physical Therapy (PT) for Veterans With Knee Osteoarthritis (Group PT): Function QUERI 2.0
Acronym: Group PT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 21-003; QUE 20-023 (Other Grant/Funding Number: VA Quality Enhancement Research initiative (QUERI))
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis of Knee; Functional Independence; Quality of Life; Implementation Science; Veterans; Group Physiotherapy; Physical Therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Parallel cluster-randomized trial (parallel-CRT): used in pragmatic evaluations of health program or policy interventions, where half the clusters (in this case, VA medical centers) are randomly assigned to two interventions: Foundational REP (active comparator) vs. Enhanced REP (experimental)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Foundational REP (Active Comparator): Foundational REP uses the Replicating Effective Program implementation strategy and includes 5 elements that were developed and tested in our prior Function QUERI work: Stakeholder engagement; Toolkit; SharePoint access for clinical program training materials; Data dashboard to assist sites with tracking their own data; and Diffusion Networks to promote peer-to-peer sharing and implementation support.
  Interventions: Other: Implementation Strategy: Foundational REP
- Enhanced REP (Experimental): EnREP begins with the same activities as foundational REP. Sites that do not meet EBP-specific a priori benchmarks reflecting adoption within 6 months will continue with foundational REP and will receive higher intensity support for a period of 6 months (enREP). Additionally, sites randomized to enREP that met adoption benchmarks but did do not meet the sustainment benchmark, will also receive intensified implementation support for the remainder of the study period (3 months). The higher intensity support will include one-on-one calls approximately every 3 to 4 weeks between site implementation teams and a trained practice facilitator (from Function QUERI team). The facilitator will coach individual sites using techniques, processes, and activities to help teams make decisions and identify and solve problems. Facilitators' actions will depend on each site's needs and clinical context.
  Interventions: Other: Implementation Strategy: Enhanced REP (enREP)

INTERVENTIONS:
Other: Implementation Strategy: Foundational REP — The goal is to test implementation intensification approaches for group PT sites that have not met implementation adoption benchmarks, specifically Foundational REP vs. Enhanced REP. The investigators propose that low intensity implementation support that promotes adapting Group PT for context and provides tools for ongoing evaluation (defined as foundational REP), will be sufficient for some but not all sites to successfully implement group PT as a clinical service.
  Arms: Foundational REP
Other: Implementation Strategy: Enhanced REP (enREP) — The goal is to test implementation intensification approaches for sites that have not met implementation adoption benchmarks, specifically Foundational REP vs. EnREP. The investigators posit that monitoring sites' progress and adding, for sites with low adoption, higher intensity strategies (defined as EnREP) that directly influence teams' capacity and skills to effectively self-organize and problem-solve will lead to higher implementation adoption, penetration, fidelity, and value.
  Arms: Enhanced REP

SUMMARY:
Implementing Group Physical Therapy (PT) for Veterans with Knee Osteoarthritis (OA): Function QUERI 2.0 (Group PT) aims to implement, evaluate and sustain Group PT in 16 VA sites using a type III effectiveness-implementation hybrid design framework, which will compare implementation strategies while also gathering information about the clinical intervention and related outcomes.

DETAILED DESCRIPTION:
Knee OA is a common and often disabling health condition that affects 14 million people in the US, and rates are about twice as high among Veterans than the general population. Forty-three percent of VA healthcare users report a diagnosis of arthritis (primarily OA), and of these, 63% report activity limitations due to joint symptoms. The prevalence of OA is expected to rise dramatically over the next several decades, and this will place increasing demand on the VA to provide core, evidence-based components of knee OA care, including PT. Many of the negative effects of knee OA can be successfully mitigated through PT, a recommended core component of treatment; however, many VA healthcare users with knee OA do not receive PT, and a key barrier is the high demand for PT services in the VA. Therefore, it is important to implement efficient, effective models of physical therapy care delivery for Veterans with knee OA.

Group PT for knee osteoarthritis (OA) is a 6-session group outpatient program developed by an interdisciplinary team of investigators, clinicians and administrators at the Durham VA and funded by the VA Quality Enhancement Research Initiative (QUE 20-023). In a previously conducted (at the Durham VA) randomized controlled trial (RCT) comparing group-based PT vs. traditional individual PT for knee OA, group PT resulted in equivalent or greater improvements in pain and functional outcomes compared with individual PT. This is important because the group-based model provides care to more Veterans with fewer staffing resources, thereby increasing access and efficiency.

In this trial, the investigators plan to implement the group PT clinical program at a minimum of 16 VA medical centers using a type III effectiveness-implementation hybrid design framework ,with sites enrolled and randomized to receive standard implementation support (foundational Replicating Effective Programs or foundational REP) or a higher-intensity implementation support (enhanced REP), including additional facilitation, self-organization, and team building support for sites that do not meet adoption goals at 6 months or sustainment goals at 9 months.

Objectives. The investigators plan to develop scalable approaches to implement and sustain Group PT as well as evaluate implementation with foundational REP versus the enhanced-implementation strategy (enhanced REP).

Methodology. To evaluate implementation, the investigators will randomize sites 1:1 to either foundational REP or enhanced REP (enREP). The investigators will use generalized linear models to examine the effect of foundational vs. enhanced REP on implementation outcomes at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Participating sites must meet the following criteria: 1) Clinical personnel on staff to conduct initial evaluations and lead group classes (e,g, physical therapist, PT assistant, kinesiotherapist): this should include at least 1 primary person and 1 back-up person to cover all aspects of program delivery, 2) Offer outpatient PT service, 3) Space to conduct group sessions (if implementing in-person Group PT classes), and (4) Submission of a signed participation agreement.

  * Enrolled sites will all be exposed to Foundational REP.
  * Sites not meeting benchmarks for adoption or sustainment of Group PT will receive higher-intensity implementation support (Enhanced REP).
* The clinical outcomes assessment will include all patients enrolled in Group PT that meet inclusion criteria (clinical diagnosis of knee OA).

Exclusion Criteria:

* The one Group PT site that previously participated in Function QUERI (ClinicalTrials.gov Identifier: NCT01058304) will be excluded from enrollment in this study.
* Sites that are currently offering a group class specifically for knee OA will not be eligible to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Dominick Allen, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC; Courtney H Van Houtven, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC; Susan N. Hastings, MD MHSc, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be available upon request. Prior to distribution, a local privacy officer and study statistician will certify that the dataset contains no protected health information (PHI). Data will be provided to requestor in electronic format.
  Sufficient data and descriptors will be made available to duplicate statistical analysis and confirm conclusions in publication.
  No data or statistical code that could lead to re-identification of individuals will be released.
  Data will be stored & maintained in an approved, secured location as described in the VA Research Data Inventory Form.
  The study statistician will create de-identified, publication-specific datasets that includes all variables presented in the study publication.
  Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re-identify any individual whose data are included in the dataset.
Time Frame: Available upon request
Access Criteria: Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re- identify any individual whose data are included in the dataset.

REFERENCES:
- [Derived] Allen KD, Webb S, Coffman CJ, Anderson L, Cummin G, Drake C, Tucker M, Webster A, Sperber N, Zullig LL, Hughes JM, Ballengee LA, Abbate LM, Hoenig H, Fullenkamp N, Van Houtven CH, Hastings SN. Implementation of Group Physical Therapy for Knee Osteoarthritis: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2025 Oct 1;8(10):e2535038. doi: 10.1001/jamanetworkopen.2025.35038. PMID 41037266
- [Derived] Webb S, Drake C, Coffman CJ, Sullivan C, Sperber N, Tucker M, Zullig LL, Hughes JM, Kaufman BG, Pura JA, Anderson L, Hastings SN, Van Houtven CH, Abbate LM, Hoenig H, Ballengee LA, Wang V, Allen KD. Group physical therapy for knee osteoarthritis: protocol for a hybrid type III effectiveness-implementation trial. Implement Sci Commun. 2023 Oct 12;4(1):125. doi: 10.1186/s43058-023-00502-7. PMID 37828564
- [Derived] Hughes JM, Zullig LL, Choate AL, Decosimo KP, Wang V, Van Houtven CH, Allen KD, Nicole Hastings S. Intensification of Implementation Strategies: Developing a Model of Foundational and Enhanced Implementation Approaches to Support National Adoption and Scale-up. Gerontologist. 2023 Mar 21;63(3):604-613. doi: 10.1093/geront/gnac130. PMID 36029028
- See also: Durham VA Optimizing Function and Independence QUERI — https://www.durham.hsrd.research.va.gov/Function_Independence_QUERI.asp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: VA facilities (medical centers, community based outpatient clinics, and smaller clinics) were enrolled in three successive cohorts from June 2021 to February 2023.
Units Other Than Participants: VA Facilities
Groups:
- Foundational REP: Foundational REP uses the Replicating Effective Program implementation strategy and includes 5 elements that were developed and tested in our prior Function QUERI work: Stakeholder engagement; Toolkit; SharePoint access for clinical program training materials; Data dashboard to assist sites with tracking their own data; and Diffusion Networks to promote peer-to-peer sharing and implementation support.
  Implementation Strategy: Foundational REP: The goal is to test implementation intensification approaches for Group PT sites that have not met implementation adoption benchmarks, specifically Foundational REP vs. Enhanced REP (EnREP). The investigators propose that low intensity implementation support that promotes adapting Group PT for context and provides tools for ongoing evaluation (defined as foundational REP), will be sufficient for some but not all sites to successfully implement group PT as a clinical service.
- Enhanced REP: EnREP begins with the same activities as foundational REP. Sites that do not meet EBP-specific a priori benchmarks reflecting adoption within 6 months will continue with foundational REP and will receive higher intensity support for a period of 6 months (enREP). Additionally, sites randomized to enREP that met adoption benchmarks but did do not meet the sustainment benchmark at 9 months, will also receive intensified implementation support for the remainder of the study period (3 months). The higher intensity support will include one-on-one calls approximately every 3 to 4 weeks between site implementation teams and a trained practice facilitator (from Function QUERI team). The facilitator will coach individual sites using techniques, processes, and activities to help teams make decisions and identify and solve problems. Facilitators' actions will depend on each site's needs and clinical context.
  Implementation Strategy: Enhanced REP (enREP): The goal is to test implementation intensification approaches for sites that have not met implementation adoption benchmarks, specifically Foundational REP vs. EnREP. The investigators posit that monitoring sites' progress and adding higher intensity strategies, for sites not meeting program benchmarks (defined as EnREP), which directly influence teams' capacity and skills to effectively self-organize and problem-solve, will lead to higher implementation adoption, penetration, fidelity, and value.
Period: Overall Study
Arm/Group | Foundational REP | Enhanced REP
Started | NA; 9 VA Facilities (Data were collected at the site level. The unit of analysis for this study is VA facilities.) | NA; 10 VA Facilities (Data were collected at the site level. The unit of analysis for this study is VA facilities.)
Completed | NA; 9 VA Facilities (Data were collected at the site level. The unit of analysis for this study is VA facilities.) | NA; 9 VA Facilities (Data were collected at the site level. The unit of analysis for this study is VA facilities.)
Not Completed | NA; 0 VA Facilities | NA; 1 VA Facilities

BASELINE CHARACTERISTICS:
Population: Data were collected at the site level. The unit of analysis for this study is VA facilities.
Units Other Than Participants: VA Facilities
Groups:
- Total: Total of all reporting groups
Arm/Group | Foundational REP | Enhanced REP | Total
Number analyzed (Participants) | NA | NA | NA
Number analyzed (VA Facilities) | 9 | 10 | 19
Age, Customized [Count of Units; unit: VA Facilities] | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Units; unit: VA Facilities] — Population: Data was collected at the site level and these characteristics were not relevant and not collected.
  VA Facilities
    number analyzed (VA Facilities) | 0 | 0 | 0
    Female |  |  | 0
    Male |  |  | 0
Ethnicity (NIH/OMB) [Count of Units; unit: VA Facilities]
  Hispanic or Latino | NA — Data was collected at the site level and these characteristics were not relevant and not collected | NA — Data was collected at the site level and these characteristics were not relevant and not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Not Hispanic or Latino | NA — Data was collected at the site level and these characteristics were not relevant and not collected | NA — Data was collected at the site level and these characteristics were not relevant and not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — Data was collected at the site level and these characteristics were not relevant and not collected | NA — Data was collected at the site level and these characteristics were not relevant and not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Count of Units; unit: VA Facilities] — Based on geographic census region.
  VA Facilities
    United States: Northeast | 2 | 2 | 4
    United States: Midwest | 0 | 2 | 2
    United States: South | 5 | 3 | 8
    United States: West | 2 | 3 | 5
Facility Complexity [Count of Units; unit: VA Facilities] — Defined using a VA facility-level measure that reflects the complexity of services offered. There are five classifications: 1a (most complex), 1b, 1c, 2, or 3 (least complex).
  VA Facilities
    High Complexity (1a) | 5 | 6 | 11
    Medium-Low Complexity (1b, 1c, 2, 3) | 4 | 4 | 8
Implementation Experience [Count of Units; unit: VA Facilities]
  Quite a lot or a fair bit | 8 | 7 | 15
  Some | 1 | 2 | 3
  Very little or none | 0 | 1 | 1
Rurality [Count of Units; unit: VA Facilities] — Determined using the VA Office of Rural Health (ORH) rurality calculator, which uses the closest facility or county/zip code to determine percent of rural Veterans served. We dichotomized rurality as high (≥50%) and low (<50%).
  VA Facilities
    High | 1 | 3 | 4
    Low | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Penetration
Description: Penetration is defined as the average number of patients enrolling in the group physical therapy (PT) program on a monthly basis (defined as completing at least one class).
Time Frame: 7-12 months
Population: Data were collected at the site level. The unit of analysis for this study is VA facilities.
Measure: Mean (Standard Deviation); unit: patients per month
Units Other Than Participants: VA Facilities
Arm/Group | Foundational REP | Enhanced REP
Number analyzed (Participants) | NA | NA
Number analyzed (VA Facilities) | 9 | 10
patients per month | 1.41 (1.15) | 1.13 (0.94)
Statistical Analysis 1: Comparison: Foundational REP vs Enhanced REP; Models included the arm indicator variable in addition to the stratification variables used in randomization: site complexity level (high complexity '1a', '1b' or '1c' vs. all others) and rurality (high sites serving ≥50% rural/highly rural Veterans vs. low sites serving <50% rural/highly rural Veterans); Test type: Superiority; p = 0.92, Regression, Linear; Mean Difference (Net) = -0.05, 95% CI 2-sided [-1.07 to 0.98]

2. Secondary Outcome: Fidelity
Description: Fidelity will be the average number of group PT sessions attended by patients who enroll in the program.
Time Frame: 7-12 months
Population: Data were collected at the site level. The unit of analysis for this study is VA facilities. Fidelity was only relevant to patients that attended Group PT sessions; therefore, calculations only included sites that held a Group PT class (Foundational sites = 7, Enhanced sites = 9) and capped class attendance at 6 classes maximum (although sites could allow patients to attend more than 6 classes).
Measure: Mean (Standard Deviation); unit: Classes per patient
Units Other Than Participants: VA Facilities
Arm/Group | Foundational REP | Enhanced REP
Number analyzed (Participants) | NA | NA
Number analyzed (VA Facilities) | 7 | 9
Classes per patient | 4.22 (0.90) | 5.01 (0.77)
Statistical Analysis 1: Comparison: Foundational REP vs Enhanced REP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.056, Regression, Linear; Mean Difference (Net) = 0.94, 95% CI 2-sided [-0.03 to 1.90]

3. Secondary Outcome: Adoption
Description: Adoption will be defined as: 1) Delivery of Group PT as a clinical service (delivery of at least 1 Group PT class) by the VA Medical Center, and 2) Enrollment of at least 5 patients.
Time Frame: 7-12 months
Population: Data were collected at the site level. The unit of analysis for this study is VA facilities. Program adoption is a binary outcome defined as delivery of Group PT as a clinical service (delivery of at least 1 Group PT class) by the VA Medical Center, and enrollment of at least 5 patients.
Measure: Number; unit: Number of VA facilities that adopted
Units Other Than Participants: VA Facilities
Arm/Group | Foundational REP | Enhanced REP
Number analyzed (Participants) | NA | NA
Number analyzed (VA Facilities) | 9 | 10
Number of VA facilities that adopted | 6 | 6

ADVERSE EVENTS:
Time Frame: Analysis was at the site level and there were no possible adverse events.
Description: All cause mortality and/or serious adverse or other (Not Including Serious) adverse events were not collected on Veterans, caregivers, or providers.
Arm/Group | Foundational REP | Enhanced REP
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT05282927/Prot_SAP_000.pdf